CLINICAL TRIAL: NCT01642394
Title: Impact of Self-care Education Program "Active Patient" in Metabolic Control, Cardiovascular Risk and Quality of Life in Patients With Type 2 Diabetes in Primary Care in the Basque Country: Randomized Clinical Trial of 2 Years of Follow up
Brief Title: Impact of Self-care Education Program in Patients With Type 2 Diabetes in Primary Care in the Basque Country
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osakidetza (Other)
Collaborators: Kronikgune-- Association Centre of International Excellence in Research on Chronicity (Unknown); Department of Health Basque Government (Unknown); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Estibaliz Gamboa Moreno, Diploma of Nursing, Osakidetza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KRONIK11/036
Record Dates: First submitted 2012-05-16; First posted 2012-07-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Chronic Disease; Education; Primary Care; Self care; Self Management
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Intervention group The complete intervention consists of group sessions (8 to 15 people) lasting 2.5 hours, once a week for six weeks. These sessions are structured with the aim of enabling participants to acquire knowledge and skills related to the disease and its management, placing a strong emphasis on proactive tools to achieve healthier lifestyles (in terms of diet, physical exercise, management of emotions, and correct use of medication, among others).
  Control group Patients assigned to the control group will receive usual care for secondary prevention of DM2 in accordance with the Osakidetza primary care protocols, which are based on clinical practice guidelines.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standardized care (No Intervention): The control group will receive usual care for secondary prevention of type 2 diabetes according to usual care in Osakidetza's primary care.
- Self-management education programme (Experimental): Attendees will receive the Diabetes Self-Management Programme in spanish version (Manejo personal de la diabetes).
  Interventions: Behavioral: Diabetes Self-Management Program

INTERVENTIONS:
Behavioral: Diabetes Self-Management Program — The intervention will be performed by patients with type 2 diabetes and health professionals and it will be divided in 6 group sessions for two and a half hours each, on a weekly basis for 6 weeks. The session content includes techniques for dealing with problems in general, promotion of exercise, nutrition concepts, proper use of medication, effective communication and basic knowledge about diabetes and its complications. The sessions are supported with educational material.
  Two leaders, previously trained in the DSMP, will lead each group. The leading status (patient or health care professional) is obtained after attending a 6-week structured program of training, a successful completion of 4 days of training sessions, and taking part in a full course for patients with a proven leader.
  Other Names: Diabetes Self-Management Programme
  Arms: Self-management education programme

SUMMARY:
Main objective:To evaluate the effectiveness of the "Diabetes Self-Management Programme" (DSMP) on the metabolic control, cardiovascular risk reduction, quality of life and self-efficacy in adult patients with type 2 diabetes, compared with current standard care of patients with type 2 diabetes, in the context of Osakidetza's Primary Care network.

Secondary objectives:

* To evaluate the impact of the implementation of DSMP in the use of health services.
* To assess the impact of DSMP in the cost of treatment of the involved population.
* To evaluate the improvement in physical activity and diet patterns among the participants.
* To describe the feasibility of implementing the DSMP in the Basque Country's primary health care system Methodology: Randomized clinical trial in which patients diagnosed with type 2 diabetes aged between 18 and 80 years pertaining to 4 primary regions of the Basque country, who agree to participate in the study, will be randomly assigned to two groups: the intervention group (the DSMP programme) and the control group. The intervention will be performed by trained patients with type 2 diabetes and health professionals and it will consist in 6 group sessions of two and a half hours each, on a weekly basis with a overall duration of 6 weeks. The session content includes techniques for dealing with problems, promotion of exercise, nutrition concepts, proper use of medication, effective communication and basic knowledge about diabetes and its complications. The sessions are supported with educational material. The main outcome is the improvement of HbA1c (glycated hemoglobin) levels. Secondary outcomes are reduction of cardiovascular risk, increase of quality of life and self-efficacy. The results will be analyzed at 6, 12 and 24 months after the intervention.

Hypothesis: An educational intervention on patients with type 2 diabetes mellitus based on the program DSMP conducted by previously trained lay persons and health professionals, improve metabolic control as measured on a 0.5% decrease in Hb A1c (Clar, 2010),compared to regular health education. On the other hand, it is expected to see improvements in the quality of life for these patients. The intervention may reduce the weight and cardiovascular risk due to changes in the physical activity and diet patterns, getting to a more appropriate use of health services and medication. It is expected that changes in the variables occur 6 months after the intervention and remain over the time

DETAILED DESCRIPTION:
Background

The management of chronic diseases (CD) is a challenge for health services. The health system must provide a more efficient and coordinated care for people with CD aimed at reducing their decompensation and improving the quality of life for both the patient and his/her family. In this task, primary care (PC) plays a key role (Bengoa, 2008).

The better living conditions and the current development of health care have produced a demographic shift in population, resulting in increased life expectancy and therefore the prevalence of CD. In the Basque Country (BC), the population over 65 has increased in recent years by 25% (EUSTAT 2005). According to the BC Health Survey of 2007, prevalence of CD is increasing in our community as 83.5% of men and 86.1% of women over 65 have a chronic disease (Arcelay, 2009). In the health system, 80% of primary care consultations are caused by CD, representing 60% of hospital admissions and 70% of health spending (Bengoa, 2008).

The incidence of diabetes mellitus type 2 (DM2) in the BC has also increased in recent years. Currently, it is estimated that the prevalence of DM2 may be up to 12% in people over 30 years. An evaluation of the diabetic population coverage in primary care records estimates that up to 4% of the diabetic population remains undiagnosed.

Cardiovascular morbidity and mortality in people with DM2 is higher than in the general population. The mortality rate for diabetes is between 13 and 30 deaths per 100,000 people per year. 75% of patients with diabetes die due to cardiovascular disease, especially coronary heart disease. Between 6.3% and 7.4% of the spending in our health care system is deemed to be caused by diabetes. Self-promotion has a paramount importance in diabetes care (diabetes Strategy in the National Health System, 2007). It is estimated that 42% of diabetics in our community are obese, 79.6% are hypertensive and 22% have diabetic macroangiopathy (Arteagoitia, 2003).

The control of diabetes in our country, according to the latest assessment of the preferential offer of the BC, can be improved. 44% are well-controlled diabetic patients, i.e. A1 Hb less than 7%, and only 25% have blood pressure (BP) below 140/90.

These data contrast with those obtained in the final report of the GEDAPS (Red Group Study of Diabetes in Primary Health Care, 2010) covering the year 2007, in which the figures were 59% for HbA1c and 65,1% for BP. One of the proposals, raised by the group GEDAPS to improve control of patients, is the increase of educational activities to patients.

As in other developed countries, the health system in Spain has completed a cycle and requires a new organizational model to meet the challenge of chronic patient care (Department of Health Basque Government, 2010). There are different proposals to meet that challenge. Among the most developed and evaluated, we find the models for managing chronic diseases (Chronic Care Model) and the Pyramid Model of Risk (Bengoa, 2008). In both programs, self-care and education involving the subject's participation in the management of their disease have a critical role.

To achieve this change in the management of chronic disease, several health administrations have suggested self-management education programs by non-professionals. The most widely used and structured approach, with the greatest evidence of its effectiveness, is the Chronic Disease Self-Management Program (CDSMP) of Stanford University, which has been implemented in 12 countries, including UK´s Expert Patient Programme, Australia´s Partners in Health and Canada's Chronic Disease Self-Management Programme.

The CDSMP is based on the self-efficacy theory of Albert Bandura, a social cognitive theory, which states that the key predictors of successful change in behaviour are confidence (self-efficacy) in the ability to perform an action and the prospect of achieving a particular goal (expected outcome). Self-efficacy is considered the first step in the causal pathways of behavior change in self-care programmes. Increased self-efficacy is a prerequisite for behaviour change through an improvement in the treatment of chronic disease, resulting in lower demand for health care (Foster, 2007).

The CDSMP was designed at Stanford University in California. It was developed and evaluated for 20 years, through randomized controlled trials (Gordon, 2008). The first program was the "Course of arthritis self-management" which later became the prototype of the following courses of self-management. They have developed a specific self-management course for diabetes, "Diabetes Self-Management Programme (DSMP)", which in the Spanish version is called "Manejo Personal de la Diabetes (MPD)"

Each patient is trained through structured courses, to complete personal action plans designed to take control of his life with chronic illness. The mission of the leaders, two in each course, is to assist patients in problem solving, decision making and self-efficacy. Leaders are usually non-professionals with one or more chronic diseases, but caregivers of chronic patients could act as leaders as well

Education by non-professionals differs from education provided by professionals:

* Commonly they live with chronic illnesses so they can act as role models for participants.
* The format is less formal in order to promote discussion on ways of self care that participants consider useful, and might not feel able to discuss in a program run by professionals.
* Lay leaders, especially for certain ethnic groups, can provide a subtle but important interpretation of health advice.

Research Question

Is a self-management education programme taught by non-professionals (DSMP) for type 2 diabetes living in the Basque Country more effective than regular health education, evaluated in terms of improvement in HbA1c, quality of life, self-efficacy,cost and other clinical variables(BP, cardiovascular risk, BMI, etc)

Justification for the novelty of the question, the expected progress beyond what is currently known.

Many systematic reviews (SR) about the effectiveness of these models have been published (Foster, 2007) (Gordon, 2008) (Bury, 2005). RS conducted by Chodosh (Chodosh et al., 2005), limited to old people, found benefits in outcome variables (blood pressure and glycosylated hemoglobin) in diseases such as diabetes and hypertension but not in osteoarthritis. The Cochrane's SR (Foster, 2007) evaluated 17 clinical trials (EK), none of them taking place in our environment, and includes references that appear in the report of the NICE (Bury, 2005). Seven of the studies were on CDSMP. The diseases included were arthritis, diabetes, hypertension and chronic pain. Their conclusions differ from Chodosh's, because Cochrane's SR obtains small but significant differences in self-rated health, aerobic physical exercise and cognitive treatment of symptoms but no evidence on variables such as psychological health, quality of life or number of visits to the general practitioner.

In Spain, Andalucía (Andalusian School of Public Health) and Catalonia (Catalan Health Institute) have experience in chronic disease programmes following this model. Both cases had preliminary favourable results. However, they have not been evaluated prospectively and neither of them has been compared with usual care or with other structured programs (Gonzalez Mestre, 2009)

A very recent study, performed in another health care setting (male veterans in the U.S.), has shown that an educational intervention conducted by patients is more effective in glycemic control than educational intervention conducted by nurses (Heisler, 2010).

Another recently published study conducted in primary care in Ireland using also patients has not been shown effective in patients with type 2 diabetes. The program used is not the Chronic Disease Self-Management Programme (CDSMP) (Smith, 2011).

Although educational group interventions by health care professionals have proven effectiveness (Deakin, 2008), they are not a regular practice in Osakidetza's Primary Care

In summary, we can conclude from the literature review that:

* There are no assessments by prospective controlled studies of these interventions in our system.
* The heterogeneity in the outcomes of interventions is a fact, due to the different lengths of studies, type of interventions and populations.
* There is no long-term assessment of effectiveness of these models.
* There is an under-representation of children and men.

Publications evaluating these models suggest the following research areas:

* Patient-centered evaluation of clinical outcomes.
* Design-studies that evaluate the use of health services.
* Cost-effectiveness studies.
* Influence of the different components of interventions on outcomes.
* Qualitative research on the way that participants experience interventions.

Given the discrepancy between the findings of the various publications, such as those in the NHS, and the lack of research in our country, we reaffirm the need for research in our system.

Feasibility of the question

The health department of the BC is supporting a new management strategy for chronic patient according to the Chronic Care Model (http://cronicidad.euskadi.net). One of the cornerstones of this model is the promotion of self-care and education of the population. Following that idea, the strategy wants to promote the "Active Patient Programme ". This programme is based on the CDSMP and the DSMP.

DM2 is a chronic disease whose management is currently carried out in our community in Primary Care (PC) and in which nursing has always had a fundamental role. PC professionals in our community have broad experience in the clinical management of diabetes in both individual patient education and treatment to prevent long term complications. Nursing has an added motivation, as one of the strategic lines of the current health department is the involvement of this group in the new ways of managing chronic illness. Nurses will likely accept programs that promote these new roles.

On the other hand, implementing this programme does not require expensive new material resources or complicated infrastructure. These programs may be conducted within daily activities of our health facilities although it may be necessary to use venues outside the health system as cultural centers, neighbourhood associations, etc…

One of the strengths of the program is the simplicity of its implementation. The program is designed to be led by patients who, after specific training and receiving standardized material support, are capable of directing groups. These patients are people with chronic illness, who voluntarily offered themselves to help other patients to learn how to self manage their disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years from four primary regions of the Basque Country: Araba, Bidasoa, Ezkerraldea- Enkarterri, Ekialde, with type 2 diabetes who have agreed to participate in the "Active Patient".

Exclusion Criteria:

* Adults over 80 years or patients with mental disorder that distorts reality (schizophrenia, bipolar disorder, Alzheimer's disease, psychosis, dementia) or morbidity which can interfere with the course, like chronic patients at home.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Glycated hemoglobin | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators are going to measure the diference between basal Glycated Hemoglobin and 6,12 and 24 months Glycated Hemoglobin.

SECONDARY OUTCOMES:
Change in Cardiovascular risk | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will use the Framingham-Regicor function
Change in quality of life | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will use the ADDQoL-19
Change in self efficacy | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will use the Stanford Spanish diabetes self-efficacy survey
Change in health services utilization | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will measure the number of visits to the general practitioner and nurse, number of visits to the emergency department and number of hospitalizations
Introduction or removal of hypoglycaemic drugs | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will compare the number of hypoglycaemic drugs before and after intervention.
Introduction or removal of antiplatelet drugs | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will compare the number of antiplatelet drugs before and after intervention.
Introduction or removal of antihypertensive drugs | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will compare the number of antihypertensive drugs before and after intervention.
Introduction or removal of lipid drugs | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will compare the number of lipid drugs before and after intervention.
Change in the percentage of patients with HbA1c less than 7% | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will consider HbA1c less than 7% as good control
Change in BMI | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  BMI (Body mass index)
Change in blood pressure | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  Systolic and diastolic blood pressure (SBP and DBP)
Change in percentage of patients with SBP <140 and DBP <80 | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will measure the diference between basal percentage of patients with SBP <140 and DBP <80 and 6,12 and 24 months percentage of patients with SBP <140 and DBP <80.
Change in the value of total cholesterol | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will measure the diference between basal total cholesterol and 6,12 and 24 months total cholesterol.
Change in the value of HDL-cholesterol | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will measure the diference between basal HDL-cholesterol and 6,12 and 24 months HDL-cholesterol.
Change in physical activity | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will use the 7 day Physical Activity Recall
Change in the diet composition | Measurements will be carried out before intervention and 6, 12 and 24 months after intervention
  The investigators will use the PREDIMED study survey. And we´ll study the percentage of people who declaring eat 5 or more daily pieces of fruit and vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: Estibaliz Gamboa Moreno, Nurse, Principal Investigator — Osakidetza
Locations (1):
- Osakidetza, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamboa Moreno E, Mateo-Abad M, Ochoa de Retana Garcia L, Vrotsou K, Del Campo Pena E, Sanchez Perez A, Martinez Carazo C, Arbonies Ortiz JC, Rua Portu MA, Pinera Elorriaga K, Zenarutzabeitia Pikatza A, Urquiza Bengoa MN, Mendez Sanpedro T, Oses Portu A, Aguirre Sorondo MB, Rotaeche Del Campo R; Osakidetza Active Patient Research Group. Efficacy of a self-management education programme on patients with type 2 diabetes in primary care: A randomised controlled trial. Prim Care Diabetes. 2019 Apr;13(2):122-133. doi: 10.1016/j.pcd.2018.10.001. Epub 2018 Nov 6. PMID 30409669
- [Derived] Gamboa Moreno E, Ochoa de Retana Garcia L, Del Campo Pena ME, Sanchez Perez A, Martinez Carazo C, Arbonies Ortiz JC, Rua Portu MA, Pinera Elorriaga K, Zenarutzabeitia Pikatza A, Urquiza Bengoa MN, Mendez Sanpedro T, Oses Portu A, Gorostidi Fano L, Aguirre Sorondo MB, Vrotsou K, Rotaeche Del Campo R. A Pilot Study to Assess the Feasibility of the Spanish Diabetes Self-Management Program in the Basque Country. J Diabetes Res. 2016;2016:9145673. doi: 10.1155/2016/9145673. Epub 2016 Dec 29. PMID 28119932
- [Derived] Gamboa Moreno E, Sanchez Perez A, Vrotsou K, Arbonies Ortiz JC, Del Campo Pena E, Ochoa de Retana Garcia L, Rua Portu MA, Pinera Elorriaga K, Zenarutzabeitia Pikatza A, Urquiza Bengoa MN, Sanz Echave R, Mendez Sampedro T, Oses Portu A, Gorostidi Fano L, Aguirre Sorondo MB, Rotaeche Del Campo R; Osakidetza Active Patient Research Group. Impact of a self-care education programme on patients with type 2 diabetes in primary care in the Basque Country. BMC Public Health. 2013 May 29;13:521. doi: 10.1186/1471-2458-13-521. PMID 23718222
- See also: In this URL you can read more information about the self-management program we are using. — http://www.osakidetza.euskadi.eus/pacienteactivo/